CLINICAL TRIAL: NCT02298478
Title: Efficacy of an Internet-based Treatment for Flying Phobia: A Randomized Controlled Trial
Brief Title: Efficacy of an Internet-based Treatment for Flying Phobia: NO-FEAR Airlines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UJaumeI05
Record Dates: First submitted 2014-11-03; First posted 2014-11-24 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Flying Phobia
Keywords: Self-help; Computer-aided Treatment; Internet; Flying phobia; minimal contact therapies; Cognitive-Behavioural Treatment; Waiting list control group
MeSH Terms: conditions — Aerophobia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group without support by the therapist (Experimental): Intervention group that do the "NO-FEAR Airlines" program and does not receive support by the therapist.
  Interventions: Behavioral: NO-FEAR Airlines
- Group with support by the therapist (Experimental): Intervention group that do the "NO-FEAR Airlines" program and receives support by the therapist (a brief weekly five-minutes call).
  Interventions: Behavioral: NO-FEAR Airlines
- Waiting list control group (Other): Control group that could access the "NO-FEAR Airlines" program after waiting for 6 weeks.
  After that time, those participants still interested were randomly assigned to one of two intervention conditions (with or without support by the therapist).
  Interventions: Behavioral: NO-FEAR Airlines

INTERVENTIONS:
Behavioral: NO-FEAR Airlines — "NO-FEAR Airlines" is a computer program that allows people who are afraid to fly to be exposed to images and sounds related to their phobic fears on a standard personal computer. The treatment can be totally self-applied.
  "NO-FEAR Airlines" divides the flight process into six sequential stages: (1) flight preparation, (2) a series of activities immediately prior to flying on the day of the flight, (3) boarding and taking off, (4) the central part of the flight, (5) the airplane's descent, approach to the runway and landing, (6) sequence with images and auditory stimuli related to plane crashes.
  Other Names: SIN MIEDO Airlines; Computer-aided Self-help Treatment for Flying Phobia; Internet-based treatment for flying phobia

SUMMARY:
The purpose of this study is to determine the efficacy of a computer-aided self-help treatment for flying phobia with or without support by the therapist, compared to a waiting list control group.

Secondary objectives: a) to explore two ways of delivering NO-FEAR Airlines, with or without therapist guidance and b) to study the patients' acceptability through expectations, preferences and satisfaction towards the online program. In this work, we present the study design.

The principal hypothesis is that the two intervention groups will improve significantly compared to the waiting list control group.

DETAILED DESCRIPTION:
One of the most prevalent phobias in our society is the fear of flying or flying phobia (FP). Surveys which identify clinically significant phobias estimate point prevalence at approximately 2.5% of the adult population. Around 10% of the general population do not fly due to intense fear, 25% of the population that fly experience intense distress during the flight and 20% of people depend on alcohol or tranquilizers to overcome the fear of flying.

The most effective psychological technique for the treatment of phobias is in vivo exposure. Besides, not all patients benefit from in vivo exposure, given that an important amount of them do not accept the intervention or drop out (around 25%) when they are informed about the intervention procedure or they have problems to access to these therapies.

Information and Communication Technologies (ICT) are pioneer applications that can improve treatment adherence and acceptance. Specifically, Computerized programs boasts remarkable advantages beyond strictly therapeutic and effectiveness-related ones in treating fear of flying: a reduction in direct therapeutic contact time, the possibility of standardizing treatment to the maximum, the low cost - which allows a greater extension - and, perhaps most importantly, access to patients who would not be very willing to subject themselves to live exposure (a real flight) with a steep exposure gradient. The application of cognitive-behavioural procedures such as exposure through interactive computer programs is especially recommended.

ELIGIBILITY:
Inclusion Criteria:

* Be older than 18 years of age,
* To meet current DSM-5 criteria for specific phobia (flying phobia).
* Be willing to participate in the study.
* Be able to use a computer and having an Internet connection at home.
* Be able to understand and read Spanish.
* Have an e-mail address.

Exclusion Criteria:

* Be receiving psychological treatment for fear of flying.
* A severe mental disorder: abuse or dependence of alcohol or other substances, psychotic disorder, dementia or bipolar disorder.
* Presence of depressive symptomatology, suicidal ideation or plan.
* Presence of heart disease.
* Pregnant women (from the fourth month).

Receiving pharmacological treatment is not an exclusion criterion during the study period, but the increase, decrease and/or change in the medication during the study period will imply the participant's exclusion from subsequent analyses.

Participants with comorbid and related disorders (i.e., panic disorder, agoraphobia, claustrophobia or acrophobia) will be included once flying phobia is the primary diagnosis. In contrast, participants who do not meet inclusion criteria will be encouraged to seek treatment alternatives better suited to their specific needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The Fear of Flying Questionnaire-II (FFQ-II; Bornas, Tortella-Feliu, García de la Banda, Fullana, & Llabrés, 1999). | up to 12 months
  The FFQ is a 30-item self-report instrument describing situations related to flying: anxiety during flight, anxiety experienced getting on the plane, and anxiety experienced by the observation of neutral or unpleasant flying related situations. For each item, respondents rated their degree of discomfort associated with the situation on a scale of 1 to 9 (1 = not at all, 9 = very much). Scores ranged from 30 to 270. As reported by Bornas et al. (1999), internal consistency was α = .97 and retest reliability (15-day retest period) was r = .92.
The Fear of Flying scale (FFS; Haug et al. (1987) | up to 12 months
  FFS is a 21-item self-report measure for assessing fear associated with various air travel situations. Fear elicited by each situation was rated on a 5-point scale (0 = not at all, 4 = very much), with scores ranging from 0 to 84. In the original FFS (Haug et al., 1987) Cronbach's alpha was .94 and retest reliability (at three months) was .86.

SECONDARY OUTCOMES:
Fear and Avoidance Scales (adapted from Marks & Mathews, 1979) | up to 12 months
  Participants assessed their fear and avoidance on a scale ranging from 0 ("No fear at all," "I never avoid") to 10 ("Severe fear," "I always avoid") for situations related to flying.
  The degree of belief in catastrophic thought was also assessed on a 0 to 10 scale.
The Fear of flying scale (FFS; Haug et al., 1987) | up to 12 months
  FFS is a 21-item self-report measure for assessing fear associated with various air travel situations. Fear elicited by each situation was rated on a 5-point scale (0 = not at all, 4 = very much), with scores ranging from 0 to 84. In the original FFS (Haug et al., 1987) Cronbach's alpha was .94 and retest reliability (at three months) was .86.

OTHER OUTCOMES:
The Patient improvement Scale (Adapted from the Clinical Global Impression scale, CGI; Guy, 1976). | up to 12 months
  One item of the CGI scale was adapted in order to assess the level of improvement achieved by the patient (compared to the baseline status) on a 7-point scale (1 "much worse" to 7 "much better"). This scale is answered by the patient.
Treatment Preferences Questionnaire (Labpsitec, 2015) | up to 12 months
  This instrument was specifically developed for this research. It is composed by 5 questions to measure participant's preferences regarding both treatment conditions included in this study (with and without therapist support): (1) Preference (2) Subjective effectiveness 3) Logical (4) Subjective aversion (5) Recommendation. Questions are composed by two response options in accordance with the two treatment conditions. This scale will be completed before participants know the treatment condition assigned and after treatment.
Qualitative interview (Labpsitec, 2015). | up to 12 months
  This interview was also specifically developed for this research. It contains 11 items in order to assess participants' opinion regarding NO-FEAR Airlines program and about the support received. The interview includes questions that are rated on 1 to 5 scales (1= very little; 5= very much) and Dichotomous Questions ("Yes" or "No"). Additionally, options to extend the qualitative participants' responses are available.

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Quero, Full professor, Study Director — University Jaume I, Castellon, Spain.; Juana Bretón, Assistant professor, Study Director — University Jaume I, Castellon, Spain.; Daniel Campos, PhD student, Study Chair — University Jaume I, Castellon, Spain
Locations (1):
- University Jaume I, Castellon, Castellon, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tortella-Feliu M, Botella C, Llabres J, Breton-Lopez JM, del Amo AR, Banos RM, Gelabert JM. Virtual reality versus computer-aided exposure treatments for fear of flying. Behav Modif. 2011 Jan;35(1):3-30. doi: 10.1177/0145445510390801. PMID 21177516
- [Background] Bornas, X., Fullana, M.A., Tortella-Feliu, M., Llabrés, J. & García de la Banda, G. Computer-assisted therapy in the treatment of flight phobia: a case report. Cognitive and Behavioral Practice, 8, 234-240, 2001.
- [Background] Bornas, X., Tortella-Feliu, M. & Llabrés, J. Do all treatments work for flight phobia? Computer-assisted exposure versus a brief multicomponent nonexposure treatment. Psychotherapy Research, 16, 41-50, 2006.
- [Background] Bornas, X., Tortella-Feliu, M., García de la Banda, G., Fullana, M. A., & Llabrés, J. Validación factorial del Cuestionario de Miedo a Volar [Factorial validation of the Fear of Flying Questionnaire]. Análisis y Modificación de Conducta, 25, 885-907, 1999.
- [Background] Botella C, Quero S, Banos RM, Garcia-Palacios A, Breton-Lopez J, Alcaniz M, Fabregat S. Telepsychology and self-help: the treatment of phobias using the internet. Cyberpsychol Behav. 2008 Dec;11(6):659-64. doi: 10.1089/cpb.2008.0012. PMID 18991528
- [Background] Quero S, Campos D, Riera Del Amo A, Breton-Lopez J, Tortella-Feliu M, Banos RM, Botella C. NO-FEAR Airlines: A Computer-aided Self-help Treatment for Flying Phobia. Stud Health Technol Inform. 2015;219:197-201. PMID 26799907
- [Derived] Campos D, Breton-Lopez J, Botella C, Mira A, Castilla D, Mor S, Banos R, Quero S. Efficacy of an internet-based exposure treatment for flying phobia (NO-FEAR Airlines) with and without therapist guidance: a randomized controlled trial. BMC Psychiatry. 2019 Mar 6;19(1):86. doi: 10.1186/s12888-019-2060-4. PMID 30841930
- [Derived] Campos D, Breton-Lopez J, Botella C, Mira A, Castilla D, Banos R, Tortella-Feliu M, Quero S. An Internet-based treatment for flying phobia (NO-FEAR Airlines): study protocol for a randomized controlled trial. BMC Psychiatry. 2016 Aug 20;16:296. doi: 10.1186/s12888-016-0996-1. PMID 27544428
- See also: Laboratory of Psychology and Technology of the University Jaume I (Labpsitec) — http://www.labpsitec.uji.es
- See also: NO-FEAR Airlines website — http://www.fobiavolar.es/